CLINICAL TRIAL: NCT05096988
Title: A Study to Evaluate the Acceptability, Tolerance and Adherence of Children and Adults Consuming PKU Sphere Liquid, a Food for Special Medical Purposes (FSMP), for the Dietary Management of Phenylketonuria (PKU)
Brief Title: Evaluation of PKU Sphere Liquid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-GMPL-2018-02-21; 271801 (Other: IRAS); 20/NW/0273 (Other: HRA)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonurias
Keywords: PKU; Sphere; Liquid
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKU sphere liquid (Experimental): PKU sphere liquid will be prescribed by the study dietitian based on the patient's individual requirements.
  Interventions: Dietary Supplement: PKU sphere liquid

INTERVENTIONS:
Dietary Supplement: PKU sphere liquid — PKU sphere liquid will be prescribed by the study dietitian based on the patient's individual requirements.

SUMMARY:
PKU Sphere Liquid is a prospective, open-label, acceptability study to evaluate PKU sphere liquid in up to 15 participants aged 3 and above for the dietary management of PKU over 31 days.

DETAILED DESCRIPTION:
PKU Sphere Liquid is a newly-developed Food for Special Medical Purposes (FSMP) designed for the dietary management of patients with phenylketonuria (PKU).

PKU sphere liquid is a vanilla flavoured, ready-to-drink, low phenylalanine protein substitute containing a blend of casein glycomacropeptide (GMP) isolate, essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals, and Docosachexaenoic acid (DHA).

This is a feasibility study designed to evaluate the acceptability, tolerance and adherence of children and adults consuming PKU sphere liquid.

Participants will be given a four-week supply of PKU Sphere Liquid and they will be asked to complete a daily diary and short questionnaire for four weeks to record information on: adherence, gastrointestinal tolerance, palatability and how the product is used.

Each participant will be on the trial for 31 days. This includes a 3-day baseline period and 28 days taking the study product. If deemed appropriate in each individual circumstance, the sponsor of the trial, Vitaflo International Ltd, will continue to supply the product free of charge at the end of the trial until available on prescription.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU requiring a low protein diet and protein substitute.
* Aged three (3) years and over
* Already taking a minimum of one GMP based protein substitute per day or have previously taken one
* Able to comply with the study protocol and take the study product, according to the opinion of the PI.
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator.
* Any co-morbidity, which, in the opinion of the investigator, would preclude participation in the study.
* Diagnosis of persistent hyperphenylalaninaemia, or mild PKU not requiring dietary intervention with a low protein diet and protein supplement.
* Unwilling/unable to take a GMP based protein substitute.
* Women who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study period.

N.B.: Women who become pregnant unexpectedly during this study will be immediately withdrawn from the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Questionnaire of self-reported adherence to the prescribed amount of study product | 4 weeks
  Assessment of participant's adherence to prescribed amount during the eight week intake of the study product
Product acceptability rated on a Likert scale by the participant after four week intake | 4 weeks
  Assessment of participant's acceptability following four week intake of the study product Scale is from 1 to 5: 1 = Loved it, 5 = Really didn't like it
Questionnaire of self-reported changes in gastrointestinal tolerance during four week intake | 4 weeks
  Assessment of participant's gastrointestinal tolerance during the four week intake of the study product

CONTACTS AND LOCATIONS:
Overall Officials: Anita Macdonald, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Royal Victoria Hospital, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No